CLINICAL TRIAL: NCT05991154
Title: Increasing Access to Mental Health Support for 18-25 Year Old Indigenous Youth With the JoyPop Mobile Mental Health App: Randomized Controlled Trial
Brief Title: JoyPop Mobile Mental Health App With Indigenous Transitional-Aged Youth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lakehead University (Other)
Collaborators: Dilico Anishinabek Family Care (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 100157(1)
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Emotion Regulation; Depression; Anxiety; Stress
Keywords: eHealth; mobile health; smartphone; emotion regulation; Indigenous; First Nations; mental health; youth; transitional-aged youth; waitlist
MeSH Terms: conditions — Emotional Regulation; Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: A pragmatic, parallel arm randomized controlled superiority trial will be used. Participants will be randomly allocated in a 1:1 ratio to the control (usual practice; UP) or intervention (UP + JoyPop) condition. Stratified block randomization (block size of 10) will be used to randomly assign participants to each condition.
Who Masked: Investigator
Masking Description: Given the nature of this trial, it will not be possible to blind participants to their allocation. As measures are self-report, blinding of outcome measures is also not possible. Protect against bias will occur by blinding investigators to condition (i.e., only staff directly managing participants will be unblinded).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Practice + JoyPop (Experimental): Participants will be monitored through the existing wait-list practices, which involve regular phone calls to check in and assess functioning, and will receive access to the JoyPop app for 4 weeks.
  Interventions: Behavioral: Usual Practice + JoyPop
- Usual Practice (No Intervention): Participants will be monitored through existing wait-list practices which involve regular phone calls to check in and assess functioning. After 4 weeks in the Usual Practice condition, participants will be offered access to the JoyPop app.

INTERVENTIONS:
Behavioral: Usual Practice + JoyPop — Participants will be asked to use the app at least twice daily but will otherwise not be provided with requirements related to feature or total usage.
  Arms: Usual Practice + JoyPop

SUMMARY:
Indigenous youth in Northwestern Ontario who need mental health supports experience longer waits than non-Indigenous youth within the region and when compared to youth in other more urban areas. Limited access and extended waits can exacerbate symptoms, prolong distress, and increase risk for more serious outcomes. Transitional aged youth (i.e., those in their mid-late teens to early twenties) are a particularly vulnerable group. Novel, innovative approaches are urgently needed to provide support for Indigenous youth in Northwestern Ontario. In partnership with Dilico Anishinabek Family Care, the investigators are evaluating the impact of a mental health app (JoyPop) as a tool for Indigenous transitional-aged youth who are waiting for mental health services. The JoyPop app was developed to support improved emotion regulation - a key difficulty for youth presenting with mental health challenges. A two-arm randomized controlled trial (RCT) will be used to evaluate the effectiveness of the app compared to usual practice while Indigenous transitional-aged youth are waiting for mental health services.

DETAILED DESCRIPTION:
Indigenous youth in Northwestern Ontario who need mental health supports experience longer waits than non-Indigenous youth within the region and when compared to youth in other more urban areas. Limited access and extended waits can exacerbate symptoms, prolong distress, increase risk for more serious outcomes like suicide, self-harm, and hospitalization, and negatively impact engagement in treatment once it is offered. Transitional aged youth (i.e., those in their mid-late teens to early twenties) are a particularly vulnerable group as they are navigating many developmental challenges (e.g., identity, relationships, schooling, housing) with the loss of supports and structures that may have been in place during childhood and adolescence. Transitional aged youth in underserviced areas such as Northwestern Ontario have increased need for and decreased access to mental health treatment, especially those in rural and remote areas. Novel, innovative approaches are urgently needed to provide support for Indigenous youth in Northwestern Ontario.

In partnership with Dilico Anishinabek Family Care, the investigators are evaluating the impact of a mental health app (JoyPop) as a tool for Indigenous transitional-aged youth who are waiting for mental health services. The JoyPop app was developed to support improved emotion regulation - a key difficulty for youth presenting with mental health challenges. Despite the promise of mobile mental health apps, significant gaps exist between the growing number of apps available in the public domain and empirical demonstration of the beneficial impacts of apps for users. Of the apps that address emotion regulation, most have not been evaluated, are narrow in scope, or have only been evaluated among non-diverse adult populations. The JoyPop app includes a broader focus, and this research is unique given its focus on rigorously evaluating the JoyPop app as a tool for treatment-seeking, Indigenous transitional-aged youth in Northwestern Ontario.

Using a randomized controlled trial (RCT) design, the primary objective is to determine the effectiveness of the JoyPop app in improving emotion regulation among Indigenous transitional-aged youth (18-25) who are waiting for mental health services as compared to usual practice (UP; monitoring those on the wait-list). The secondary objectives are to: (1) Assess change in mental health difficulties and treatment readiness between youth in each condition to better understand the app's broader impact as a wait-list tool; (2) Conduct an economic analysis to determine whether receiving the app while waiting for mental health services reduces other health service use and associated costs; (3) Define the Minimal Clinically Important Difference (MCID) for the primary outcome measure; and (4) Assess youth perspective the quality of the JoyPop app.

ELIGIBILITY:
Inclusion Criteria:

* Indigenous transitional-aged youth must be on the wait-list for mental health services at Dilico Anishinabek Family Care and be between 18-25 years old.
* Eligible youth will also need to be available to attend a virtual or in-person orientation session.
* In order to download the JoyPop app, participants will need access to an iOS device (e.g., iPhone, iPad). Refurbished iPhones containing just the JoyPop app will be provided to participants to use for the duration of the trial if they do not have access to their own.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-08-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in emotion regulation (overall) | Difficulties in Emotion Regulation Scale - Short Form will be administered at baseline (pre), after 2 weeks (mid), and after 4 weeks (post)
  Emotion regulation will be assessed with the Difficulties in Emotion Regulation Scale - Short Form. Total scores range from 18 to 90 with higher scores indicating greater difficulties in emotion regulation.
Change in emotion regulation (strategies) | Difficulties in Emotion Regulation Scale - Short Form will be administered at baseline (pre), after 2 weeks (mid), and after 4 weeks (post)
  Emotion regulation strategies will be assessed with the Difficulties in Emotion Regulation Scale - Short Form strategies subscale. Total scores range from 3 to 15 with higher scores indicating greater difficulties.
Change in emotion regulation (non-acceptance) | Difficulties in Emotion Regulation Scale - Short Form will be administered at baseline (pre), after 2 weeks (mid), and after 4 weeks (post)
  Emotion regulation strategies will be assessed with the Difficulties in Emotion Regulation Scale - Short Form non-acceptance subscale. Total scores range from 3 to 15 with higher scores indicating greater difficulties.
Change in emotion regulation (impulse) | Difficulties in Emotion Regulation Scale - Short Form will be administered at baseline (pre), after 2 weeks (mid), and after 4 weeks (post)
  Emotion regulation strategies will be assessed with the Difficulties in Emotion Regulation Scale - Short Form impulse subscale. Total scores range from 3 to 15 with higher scores indicating greater difficulties.
Change in emotion regulation (goals) | Difficulties in Emotion Regulation Scale - Short Form will be administered at baseline (pre), after 2 weeks (mid), and after 4 weeks (post)
  Emotion regulation strategies will be assessed with the Difficulties in Emotion Regulation Scale - Short Form goals subscale. Total scores range from 3 to 15 with higher scores indicating greater difficulties.
Change in emotion regulation (awareness) | Difficulties in Emotion Regulation Scale - Short Form will be administered at baseline (pre), after 2 weeks (mid), and after 4 weeks (post)
  Emotion regulation strategies will be assessed with the Difficulties in Emotion Regulation Scale - Short Form awareness subscale. Total scores range from 3 to 15 with higher scores indicating greater difficulties.
Change in emotion regulation (clarity) | Difficulties in Emotion Regulation Scale - Short Form will be administered at baseline (pre), after 2 weeks (mid), and after 4 weeks (post)
  Emotion regulation strategies will be assessed with the Difficulties in Emotion Regulation Scale - Short Form clarity subscale. Total scores range from 3 to 15 with higher scores indicating greater difficulties.

SECONDARY OUTCOMES:
Change in psychological distress | Depression Anxiety and Stress Scale 21 will be administered at baseline (pre), after 2 weeks (mid), and after 4 weeks (post)
  Psychological distress will be assessed with the total score for all items on the Depression Anxiety and Stress Scale 21. Total scores range from 0 to 63 with higher scores indicating greater psychological distress.
Change in depressive symptoms | Depression Anxiety and Stress Scale 21 will be administered at baseline (pre), after 2 weeks (mid), and after 4 weeks (post)
  Depressive symptoms will be assessed with the Depression subscale of the Depression Anxiety and Stress Scale 21. Total scores range from 0 to 21 with higher scores indicating greater depressive symptoms.
Change in anxious symptoms | Depression Anxiety and Stress Scale 21 will be administered at baseline (pre), after 2 weeks (mid), and after 4 weeks (post)
  Depressive symptoms will be assessed with the Anxiety subscale of the Depression Anxiety and Stress Scale 21. Total scores range from 0 to 21 with higher scores indicating greater depressive symptoms.
Change in stress | Depression Anxiety and Stress Scale 21 will be administered at baseline (pre), after 2 weeks (mid), and after 4 weeks (post)
  Depressive symptoms will be assessed with the Stress subscale of the Depression Anxiety and Stress Scale 21. Total scores range from 0 to 21 with higher scores indicating greater depressive symptoms.
Change is overall difficulties | Strengths and Difficulties Questionnaire will be administered at baseline (pre), after 2 weeks (mid), and after 4 weeks (post)
  Overall difficulties will be assessed with the total score from the Strengths and Difficulties Questionnaire (all subscales except prosocial). Total scores range from 0 to 40 with higher scores indicating worse difficulties.
Change is emotional problems | Strengths and Difficulties Questionnaire will be administered at baseline (pre), after 2 weeks (mid), and after 4 weeks (post)
  Emotional problems will be assessed with the Emotional Problems subscale from the Strengths and Difficulties Questionnaire. Total scores range from 0 to 10 with higher scores indicating worse emotional problems.
Change is conduct problems | Strengths and Difficulties Questionnaire will be administered at baseline (pre), after 2 weeks (mid), and after 4 weeks (post)
  Emotional problems will be assessed with the Conduct Problems subscale from the Strengths and Difficulties Questionnaire. Total scores range from 0 to 10 with higher scores indicating worse conduct problems.
Change is hyperactivity | Strengths and Difficulties Questionnaire will be administered at baseline (pre), after 2 weeks (mid), and after 4 weeks (post)
  Emotional problems will be assessed with the Hyperactivity subscale from the Strengths and Difficulties Questionnaire. Total scores range from 0 to 10 with higher scores indicating worse hyperactivity.
Change is peer problems | Strengths and Difficulties Questionnaire will be administered at baseline (pre), after 2 weeks (mid), and after 4 weeks (post)
  Emotional problems will be assessed with the Peer Problems subscale from the Strengths and Difficulties Questionnaire. Total scores range from 0 to 10 with higher scores indicating worse peer problems.
Change is prosocial behaviour | Strengths and Difficulties Questionnaire will be administered at baseline (pre), after 2 weeks (mid), and after 4 weeks (post)
  Emotional problems will be assessed with the Prosocial subscale from the Strengths and Difficulties Questionnaire. Total scores range from 0 to 10 with higher scores indicating worse prosocial behaviour.
Change in treatment readiness | Treatment Readiness subscale of the Motivation for Youth's Treatment Scale will be administered at baseline (pre), after 2 weeks (mid), and after 4 weeks (post)
  Treatment readiness will be assessed with the Treatment Readiness subscale of the Motivation for Youth's Treatment Scale. Total scores range from 4 to 20 with higher scores indicating greater readiness.

OTHER OUTCOMES:
App quality (overall) | User Version of the Mobile Application Rating Scale will be administered to the intervention group after 4 weeks (post)
  App quality (overall) will be assessed with the User Version of the Mobile Application Rating Scale. Total scores range from 1 to 5 with higher scores indicating greater quality.
App quality (engagement) | User Version of the Mobile Application Rating Scale will be administered to the intervention group after 4 weeks (post)
  App quality (engagement) will be assessed with the Engagement subscale of the User Version of the Mobile Application Rating Scale. Total scores range from 1 to 5 with higher scores indicating greater quality (engagement).
App quality (functionality) | User Version of the Mobile Application Rating Scale will be administered to the intervention group after 4 weeks (post)
  App quality (functionality) will be assessed with the Functionality subscale of the User Version of the Mobile Application Rating Scale. Total scores range from 1 to 5 with higher scores indicating greater quality (functionality).
App quality (aesthetics) | User Version of the Mobile Application Rating Scale will be administered to the intervention group after 4 weeks (post)
  App quality (aesthetics) will be assessed with the Aesthetics subscale of the User Version of the Mobile Application Rating Scale. Total scores range from 1 to 5 with higher scores indicating greater quality (aesthetics).
App quality (information) | User Version of the Mobile Application Rating Scale will be administered to the intervention group after 4 weeks (post)
  App quality (information) will be assessed with the Information subscale of the User Version of the Mobile Application Rating Scale. Total scores range from 1 to 5 with higher scores indicating greater quality (information).
App quality (subjective) | User Version of the Mobile Application Rating Scale will be administered to the intervention group after 4 weeks (post)
  App quality (subjective) will be assessed with the Subjective subscale of the User Version of the Mobile Application Rating Scale. Total scores range from 1 to 5 with higher scores indicating greater quality (subjective).
App quality (perceived impact) | User Version of the Mobile Application Rating Scale will be administered to the intervention group after 4 weeks (post)
  App quality (perceived impact) will be assessed with the Perceived Impact subscale of the User Version of the Mobile Application Rating Scale. Total scores range from 1 to 5 with higher scores indicating greater quality (perceived impact).
Service utilization | Service utilization measure will be administered at baseline (pre), after 2 weeks (mid), and after 4 weeks (post)
  Service utilization will be assessed with 5 items asking about frequency of healthcare services accessed over the prior 2 weeks. Response options are open-ended and will be analyzed individually and as a total score across service types.
Minimal Clinically Important Difference (MCID) | GRC will be administered to the intervention group after 2 weeks (mid) and 4 weeks (post)
  On the Global Rating of Change (GRC), the smallest change in emotion regulation that participants identify as important after completing the trial will be used to calculate the MCID. The GRC is an 11-point Likert scale (ranging from -5 to +5; -5 very much worse, 0 unchanged, +5 very much better) used to indicate the degree to which emotion regulation changed for the better, for the worse, or no change after receiving the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Aislin R Mushquash, Ph.D., Principal Investigator — Lakehead University
Locations (1):
- Lakehead University, Thunder Bay, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
In accordance with the Ownership, Control, Access, and Possession (OCAPTM) standards set by the First Nations Information Governance Centre, data obtained from Indigenous youth will be owned, controlled, and managed through the partner organization Dilico Anishinabek Family Care.

REFERENCES:
- [Derived] MacIsaac A, Neufeld T, Malik I, Toombs E, Olthuis JV, Schmidt F, Dunning C, Stasiuk K, Bobinski T, Ohinmaa A, Stewart SH, Newton AS, Mushquash AR. Increasing Access to Mental Health Supports for 18- to 25-Year-Old Indigenous Youth With the JoyPop Mobile Mental Health App: Study Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Jan 30;14:e64745. doi: 10.2196/64745. PMID 39883939